CLINICAL TRIAL: NCT02001402
Title: Chinese Health Investigation of Nurse Aging
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Bai Wen-Pei (Other)
Responsible Party: Sponsor-Investigator, Bai Wen-Pei, professor, Peking University First Hospital
Organization: Peking University First Hospital (Other)
Other Study IDs: 83573214
Record Dates: First submitted 2013-11-20; First posted 2013-12-04 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-11

CONDITIONS: Lipid Depletion; Excessive Physical Exercise, Unspecified; Menopausal Syndrome
Keywords: climacteric symptoms ; nurse ;; intervention;follow-up

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A follow-up intervention for the climacteric symptoms of nurses in Peking

DETAILED DESCRIPTION:
As we all know,hormone replacement therapy (HRT) is the main therapy to climacteric symptoms.But HRT has also some disadvantages including breast cancer,cardiovascular disease and so on, especially long period of HRT. It makes us to find the non-hormone therapy. So we want to investigate the exercise on the effect of climacteric symptoms.Doing exercise is helpful for avoiding and treating many disease,including climacteric symptoms.In our previous research,we found that playing exercise can treat moderate climacteric symptoms.

ELIGIBILITY:
Inclusion Criteria:

* they are nurse ,aged40-55, lived in peking ,who are among perimenopausal women.

Exclusion Criteria:

-

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: About 2000 nurese aged 40-55 living in peking will be investigated.We will measure the symptoms of perimenopausal syndrome by kupperman index、HRQOL（health -related quality of life) to evaluate the severity of menopausal syndrome and quality of life.We choose nurses whose KMI is above 15 and divided them into intervention group and control group.In intervention group,we give them health education and exercise intervention.
Sampling Method: Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2008-08; Primary Completion 2015-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
the number of KMI | up to 2 years
  KMI is the short of Kupperman index, which is a questionnaire that assesses the severity of women's climacteric symptoms.

SECONDARY OUTCOMES:
blood lipid | up to 2 years
  blood lipid is an index to measure the effect of exercise.